CLINICAL TRIAL: NCT04440644
Title: Validazione Italiana Dello Strumento BBI (Beaumont Behavioural Inventory) Per la Valutazione Delle Alterazioni Comportamentali Nel Paziente Affetto da Malattia Del Motoneurone
Brief Title: Italian Validation of the Beaumont Behavioural Inventory (BBI)
Acronym: BBI
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: CE 2320
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; frontotemporal degeneration; behavioural changes.
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: patients with amyotrophic lateral sclerosis
  Interventions: Behavioral: BBI
- Healthy control: healthy control participants
  Interventions: Behavioral: BBI

INTERVENTIONS:
Behavioral: BBI — administration of psychometric test

SUMMARY:
Up to 50% of patients affected with amyotrophic lateral sclerosis (ALS) can show behavioral dysfunctions within the spectrum of frontotemporal degenerations (FTD) - namely, apathy, disinhibition, loss of sympathy/empathy, perseverative and stereotyped behaviours, dietary changes [Strong et al., 2017].

The Beaumont Behavioural Inventory (BBI) [Elamin et al., 2017] is a questionnaire designed for detecting FTD-spectrum behavioural changes in ALS patients. The present study aims at both validating the BBI in an Italian ALS population and determining normative cut-off values of the instrument.

ELIGIBILITY:
Inclusion Criteria:

* possible, probable or definite ALS according to El Escorial revised criteria

Exclusion Criteria:

* Any other clinically significant cardiovascular, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness that in the opinion of the investigator could interfere with the interpretation of the study results

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subject with amyotrophic lateral sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Beaumont Behavioural Inventory | 2 years
  Psychometrics

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri, Milan, Italy

REFERENCES:
- [Result] Iazzolino B, Pain D, Laura P, Aiello EN, Gallucci M, Radici A, Palumbo F, Canosa A, Moglia C, Calvo A, Mora G, Chio A. Italian adaptation of the Beaumont Behavioral Inventory (BBI): psychometric properties and clinical usability. Amyotroph Lateral Scler Frontotemporal Degener. 2022 Feb;23(1-2):81-86. doi: 10.1080/21678421.2021.1946085. Epub 2021 Jul 19. PMID 34279169